CLINICAL TRIAL: NCT04143802
Title: A Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3437943 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3437943 in Participants With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17137; J1I-MC-GZBB (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-10-28; First posted 2019-10-29 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01-15

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — retatrutide; dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3437943 (Experimental): LY3437943 administered subcutaneously (SC)
  Interventions: Drug: LY3437943
- Dulaglutide (Active Comparator): Dulaglutide administered SC
  Interventions: Drug: Dulaglutide
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3437943 — Administered SC
  Arms: LY3437943
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: Dulaglutide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn about the side effects of LY3437943 when given to participants with type 2 diabetes. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. Each enrolled participant will receive injections of LY3437943, dulaglutide, or placebo given just under the skin. For each participant, the study will last up to about 5 months and will include 16 visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Have T2DM for at least 3 months before screening and are without advanced known possible complications of diabetes mellitus
* Have a glycated hemoglobin (HbA1c) value at lead-in and screening of ≥7.0% and ≤10.5% and treated with diet and exercise alone or a stable dose of metformin for at least 3 months prior to screening
* Have had a stable body weight for the 3 months prior to randomization (<5% body weight change)
* Have a body mass index of 23 to 50 kilograms per square meter (kg/m²), inclusive
* Male participants agree to use an effective method of contraception for the duration of the study plus 90 days, which corresponds to 4 months after the last investigational product dose
* Women not of childbearing potential may participate and include those who are: infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as mullerian agenesis; or those who are postmenopausal

Exclusion Criteria:

* Have type 1 diabetes mellitus or latent autoimmune diabetes in adults
* Have uncontrolled diabetes, defined as an episode of ketoacidosis or hyperosmolar state requiring hospitalization in the 6 months prior to screening
* Have a known clinically significant gastric emptying abnormality
* Have had an episode of severe hypoglycemia
* Have a history of acute or chronic pancreatitis or fasting serum triglyceride level of >500 milligrams per deciliter (mg/dL) at screening and/or Day-2. If participant is on lipid-lowering therapies, doses must be stable for 30 days prior to screening
* Have known liver disease, obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or have elevations in aminotransferases (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) greater than 3X upper limit of normal (ULN) at screening and/or Day -2

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 106
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve of LY3437943 | Baseline through study completion (12 weeks)
  PK: AUC of LY3437943
PK: Maximum Concentration (Cmax) of LY3437943 | Baseline through study completion (12 weeks)
  PK: Cmax of LY3437943
Change from Baseline in Mean Daily Plasma Glucose (PG) | Baseline through Day 80
  Change from baseline in mean daily PG from 6-point PG profile

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Miami Research Associates, Miami, Florida
  - PRA International, Lenexa, Kansas
  - Clinical Trials of Texas, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Urva S, Coskun T, Loh MT, Du Y, Thomas MK, Gurbuz S, Haupt A, Benson CT, Hernandez-Illas M, D'Alessio DA, Milicevic Z. LY3437943, a novel triple GIP, GLP-1, and glucagon receptor agonist in people with type 2 diabetes: a phase 1b, multicentre, double-blind, placebo-controlled, randomised, multiple-ascending dose trial. Lancet. 2022 Nov 26;400(10366):1869-1881. doi: 10.1016/S0140-6736(22)02033-5. Epub 2022 Oct 27. PMID 36354040
- See also: Related Info — https://www.lillytrialguide.com/en-US/studies/adult-type-2-diabetes/GZBB#?postal=